CLINICAL TRIAL: NCT05479604
Title: Treatment of Sinus Headache Using a Novel Device That Combines Acoustic Vibration With Oscillating Expiratory Pressure: Randomized Controlled Trial
Brief Title: Treatment of Sinus Headache Using a Novel Device That Combines Acoustic Vibration With Oscillating Expiratory Pressure
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: participant non-compliance
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Amar Miglani, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-001904
Record Dates: First submitted 2022-07-27; First posted 2022-07-29 (Actual); Results first posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Facial Pain
Keywords: Facial Pressure
MeSH Terms: conditions — Facial Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- SinuSonic Group (Experimental): Subjects will use the SinuSonic device for 2 minutes twice daily for 8 weeks
  Interventions: Device: SinuSonic
- Sham Group (Sham Comparator): Subjects will use the sham device for 2 minutes twice daily for 8 weeks
  Interventions: Device: Sham Device

INTERVENTIONS:
Device: SinuSonic — Handheld device that utilizes sound and pressure combined with normal breathing to relieve nasal congestion. The device is held over the nose and creates vibrations similar to humming.
  Arms: SinuSonic Group
Device: Sham Device — Device looks exactly like study device but does not emit the same pressure or make the same noise as the study device
  Arms: Sham Group

SUMMARY:
The purpose of this study is to investigate if the SinuSonic device decreases facial pain and pressure compared to the placebo device.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be > 18 years of age inclusive, at the time of signing the informed consent.
* Participants who are overtly healthy as determined by medical evaluation including medical history and physical examination.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* Facial pain or pressure for > 3 months of symptom duration.
* Pain/pressure VAS (Visual Analogue Scale) Score of > 5.

Exclusion Criteria:

* Upper respiratory illness within the last 2 weeks.
* History of severe epistaxis.
* Known pregnancy.
* Allergic sensitivity to silicone or any other component of device.
* Sinonasal surgery in the last 3 months.
* Topical decongestant use in the last week.
* Nasal polyposis, purulence/edema, or other signs of sinusitis on exam.
* Sinusitis on imaging.
* Nasal crusting or ulceration on exam.
* Inability to read or understand English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2024-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amar Miglani, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Arizona, Phoenix, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of both pre-screening and screening measures, where screening measures took place after consent. Two participants were assigned study numbers at the time of consent and screen failed based on screening criteria. Another two participants who were assigned study numbers refused further participation following the consent visit, who met screening criteria, prior to being randomized. One participant met screening criteria, but the study was stopped prior to randomization.
Period: Overall Study
Arm/Group | SinuSonic Group | Sham Group
Started | 9 (9 Participants) | 13
Completed | 8 | 8
Not Completed | 1 | 5
Not completed — Lost to Follow-up | 1 | 5

BASELINE CHARACTERISTICS:
Population: Only complete datasets that contained all primary and secondary outcome measures at 'Baseline' and 'Week 8' timepoints were analyzed in the final data analysis process.
Groups:
- Total: Total of all reporting groups
Arm/Group | SinuSonic Group | Sham Group | Total
Number analyzed (Participants) | 9 | 13 | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52 (13.8) | 54 (11.8) | 53 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 9 | 12 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 13 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 13 | 22
Baseline Visual Analogue Scale (VAS) [Mean (Standard Deviation); unit: Units on a scale] — The Visual Analogue Scale (VAS) for Facial Pain is a validated, self-reported tool used to assess the severity of facial pain. Participants are asked to rate their current facial pain intensity on a scale from 0 to 10, with 0 indicating "no pain" and 10 representing the "worst pain imaginable." Higher scores reflect worse outcomes, meaning more severe facial pain, while lower scores indicate better outcomes, or less pain. The score is reported directly by the participant based on their subjective experience. This is a single-item measure, and no subscales or composite scores are used.
  Units on a scale | 5.8 (1.5) | 5.7 (1.9) | 5.7 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Facial Pain Visual Analogue Scale (VAS)
Description: Participants rated sinus or facial pain/pressure using a 0-10 Visual Analogue Scale (VAS) which measured the average sinus pain over the past week. The VAS was displayed as a horizontal sliding scale on an electronic survey, where participants moved a slider along a continuum from 0 = no pain to 10 = worst possible pain. The slider allowed for selection of whole-number values only. Higher scores indicate worse outcomes (greater pain); lower scores indicate better outcomes (less pain).
Time Frame: Baseline, 8 weeks
Population: Facial Pain - Visual Analogue Scale (VAS)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SinuSonic Group | Sham Group
Number analyzed (Participants) | 9 | 8
score on a scale | 2.4 (1.6) | 3.9 (2.6)

2. Primary Outcome: Change in Brief Pain Inventory Short Form (BPI-SF)
Description: The Brief Pain Inventory - Short Form (BPI-SF) is a 9-item self-report questionnaire that assesses pain severity and its impact on daily functioning. Pain intensity (worst, least, average, current) and pain interference (e.g., activity, mood, sleep) are rated on a 0-10 scale, with 0 = no pain/no interference and 10 = worst pain/completely interferes. Higher scores indicate worse outcomes, whereas lower scores indicate better outcomes.
Time Frame: Baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SinuSonic Group | Sham Group
Number analyzed (Participants) | 9 | 13
score on a scale | 2.4 (1.6) | 3.9 (2.6)

3. Secondary Outcome: Subjects Reporting Pain With Device Use
Description: Number of subjects reporting pain with device use
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | SinuSonic Group | Sham Group
Number analyzed (Participants) | 9 | 11
Participants | 0 | 0

4. Secondary Outcome: Subjects Reporting Epistaxis
Description: Number of subjects reporting epistaxis
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | SinuSonic Group | Sham Group
Number analyzed (Participants) | 9 | 11
Participants | 0 | 0

5. Secondary Outcome: Change in Nasal Obstruction Symptoms
Description: The Nasal Obstruction Symptom Evaluation (NOSE) Score is a 5-item, self-reported survey that assesses the impact of nasal obstruction on quality of life over the past month; each item is rated from 0 (not a problem) to 4 (severe problem). These five items form a single subscale (i.e., nasal obstruction symptom severity). The responses to all 5 items are summed to yield a raw total score ranging from 0 to 20. Raw scores are scaled to a total score out of 100, by multiplying by 5. Nasal Obstruction Severity Classification categories: Mild (5-25), Moderate (30-50), Severe (55-75), Extreme (80-100). A score of 0 means that there are no problems with nasal obstruction and a score of 100 means that they are experiencing the worst possible problems with nasal obstruction. NOSE scores will be obtained at 'Baseline' and 'Week 8,' to measure obstruction changes with device use (sham vs real).
Time Frame: Baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SinuSonic Group | Sham Group
Number analyzed (Participants) | 9 | 11
score on a scale | 61.1 (22.7) | 67.7 (21.9)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 8 weeks
Arm/Group | SinuSonic Group | Sham Group
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/13
Other Adverse Events (participants affected / at risk) | 1/9 | 0/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SinuSonic Group (N=9) | Sham Group (N=13)
Other specified disorders of nose and nasal sinuses (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — J34.89 - Other specified disorders of nose and nasal sinuses. Notes: patient reported nose scabbing when using the real device (not sham).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-09): https://cdn.clinicaltrials.gov/large-docs/04/NCT05479604/Prot_SAP_001.pdf